CLINICAL TRIAL: NCT05642143
Title: Deep Phenotyping of Bone Disease in Type 2 Diabetes and Relations to Diabetic Neuropathy
Status: Recruiting | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Julie Lindgård Nielsen, Principal Investigator, Aalborg University Hospital
Other Study IDs: N-20220038
Record Dates: First submitted 2022-11-04; First posted 2022-12-08 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Type 2 Diabetes; Bone Disease; Osteoporosis; Diabetic Neuropathy Peripheral; Autonomic Neuropathy, Diabetic
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Bone Diseases; Osteoporosis; Diabetic Neuropathies | interventions — Nerve Conduction Studies; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples, urine and skin biopsies
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- T2D F-/N-: Subjects with T2D and no previous history of any fractures or diabetic neuropathy (n=160)
  Interventions: Diagnostic Test: Dual Energy X-ray Absorbtiometry scan; Diagnostic Test: High-resolution peripheral quantitative computed tomography; Diagnostic Test: Microindentation; Diagnostic Test: Thermal perception thresholds; Diagnostic Test: Nerve conduction studies; Diagnostic Test: Composite Autonomic Symptom Score 31; Diagnostic Test: Skin biopsies with quantification of intra-epidermal nerve fibre density; Diagnostic Test: Perception Threshold Tracking; Diagnostic Test: Assessment of cardiovascular autonomic neuropathy; Diagnostic Test: Handgrip strength; Diagnostic Test: Force plate platform; Diagnostic Test: Biospecimen collection; Diagnostic Test: Isometric leg extension strength; Diagnostic Test: Michigan Neuropathy Screening Instrument
- T2D F+: Subjects with T2D with a previous history of a fracture(s) (any fracture, major osteoporotic fracture (MOF) and peripheral) (n=100)
  Interventions: Diagnostic Test: Dual Energy X-ray Absorbtiometry scan; Diagnostic Test: High-resolution peripheral quantitative computed tomography; Diagnostic Test: Microindentation; Diagnostic Test: Thermal perception thresholds; Diagnostic Test: Nerve conduction studies; Diagnostic Test: Composite Autonomic Symptom Score 31; Diagnostic Test: Perception Threshold Tracking; Diagnostic Test: Assessment of cardiovascular autonomic neuropathy; Diagnostic Test: Handgrip strength; Diagnostic Test: Force plate platform; Diagnostic Test: Biospecimen collection; Diagnostic Test: Isometric leg extension strength; Diagnostic Test: Michigan Neuropathy Screening Instrument
- T2D N+: Subjects with T2D matched by age and sex with severe peripheral (vibration perception threshold (VPT) > 50) or a history of autonomic neuropathy (n=40)
  Interventions: Diagnostic Test: Dual Energy X-ray Absorbtiometry scan; Diagnostic Test: High-resolution peripheral quantitative computed tomography; Diagnostic Test: Microindentation; Diagnostic Test: Thermal perception thresholds; Diagnostic Test: Nerve conduction studies; Diagnostic Test: Composite Autonomic Symptom Score 31; Diagnostic Test: Skin biopsies with quantification of intra-epidermal nerve fibre density; Diagnostic Test: Perception Threshold Tracking; Diagnostic Test: Assessment of cardiovascular autonomic neuropathy; Diagnostic Test: Handgrip strength; Diagnostic Test: Force plate platform; Diagnostic Test: Biospecimen collection; Diagnostic Test: Isometric leg extension strength; Diagnostic Test: Michigan Neuropathy Screening Instrument

INTERVENTIONS:
Diagnostic Test: Dual Energy X-ray Absorbtiometry scan — Evaluation of body composition and bone mass density
  Other Names: DXA
Diagnostic Test: High-resolution peripheral quantitative computed tomography — High-resolution peripheral quantitative computed tomography (HR-pQCT) assesses both volumetric bone mineral density (vBMD) and trabecular and cortical microarchitecture.
  Other Names: HR-pQCT
Diagnostic Test: Microindentation — Measures Bone Material Strength Index (BMSi) of cortical bone.
  Other Names: Osteoprobe, ActiveLife, Santa Barbara, CA
Diagnostic Test: Thermal perception thresholds — Heat and cold perception thresholds
  Other Names: Quantitative Sensory Testing
Diagnostic Test: Nerve conduction studies — Nerve conduction and amplitude of sural nerve
  Other Names: NCStat-DPN-Check
Diagnostic Test: Composite Autonomic Symptom Score 31 — A validated self-assessment questionnaire quantifying the severity and distribution of autonomic symptoms across six domains (orthostatic intolerance, vasomotor, secretomotor, gastrointestinal, bladder and pupillomotor functions) by scoring 31 clinically selected questions
  Other Names: COMPASS 31
Diagnostic Test: Skin biopsies with quantification of intra-epidermal nerve fibre density — Skin biopsy
  Other Names: PGP9.5, antibodies for subsets of ion-channels ect
  Groups: T2D F-/N-; T2D N+
Diagnostic Test: Perception Threshold Tracking — Transcutaneous stimulation of large and small nerve fibres using weak electrical currents
  Other Names: PTT
Diagnostic Test: Assessment of cardiovascular autonomic neuropathy — Electrocardiographic recordings at rest and during cardiovascular autonomic reflex tests.
  Other Names: Vagus device, Medicus Engineering ApS, Aarhus, Denmark
Diagnostic Test: Handgrip strength — Evaluation of muscle strength
  Other Names: Hydraulic dynamometer, Saehan Corporation, Gyungnam, South Korea
Diagnostic Test: Force plate platform — Evaluation of balance while standing still
  Other Names: Plux Biosignals, S.A, Arruda dos Vinhos, Portugal
Diagnostic Test: Biospecimen collection — Biochemistry including bone turnover markers, glycemic status, inflammation markers i.e
  Other Names: Blood samples; Urine samples
Diagnostic Test: Isometric leg extension strength — Evaluation of muscle strength
  Other Names: EasyForce Digital Dynamometer
Diagnostic Test: Michigan Neuropathy Screening Instrument — MNSI is used to assess status of peripheral neuropathy. It includes two separate assessments: a 15-item self-administered questionnaire and a lower extremity examination that includes inspection and assessment of vibratory sensation and ankle reflexes.
  Other Names: MNSI

SUMMARY:
Objectives:

The goal of this cross sectional clinical trial is to examine the phenotype of bone disease in type 2 diabetes.The main aims are to:

1. Compare bone microarchitecture, bone biomechanical competence, and bone turnover markers as well as postural control in T2D patients with and without fractures.
2. Examine how autonomic and peripheral neuropathy affects bone microarchitecture, bone material strength and bone turnover markers as well as postural control in T2D.

Methods:

The trial is of cross-sectional design and consists of examinations including

* Blood samples to analyze bone markers, glycemic state i.e.
* Bone scans including dual energy x-ray absorptiometry (DXA) and high resolution peripheral quantitative computed tomography (HRpQCT) to evaluate Bone Mineral Density, t-score and bone structure.
* Microindentation to evaluate bone material strength
* Skin autofluorescence to measure levels of advanced glycation endproducts (AGEs) in the skin
* Assesment of nerve function (peripheral and autonomic)
* Assesment of postural control, muscle strength and gait

Participants:

A total of 300 type 2 diabetes patients divided to three groups:

* 160 with no history of fractures or diabetic neuropathy
* 100 with a history of fracture(s)
* 40 with autonomic neuropathy or severe peripheral neuropathy

ELIGIBILITY:
Inclusion Criteria:

1. Men and women with minimum 40 years of age.
2. Diagnosis of T2D. At least one of the following criteria must be met at diagnosis:

   1. HbA1c ≥ 48 mmol/mol (6,5 %)
   2. Plasma glucose ≥ 11,1 mmol/l
   3. Fasting plasma glucose ≥7,0 mmol/l Clinical effect of oral antidiabetic medication strengthens the diagnosis.
3. Diagnosis of diabetes at least one year prior to inclusion of the study to avoid honeymoon diabetes.
4. A history of fracture(s) (confirmed by radiographs analyzed by radiologist) following the diabetes diagnosis (T2D F+ group)
5. Diagnosed with severe peripheral (VPT ≥ 50) or autonomic neuropathy defined by cardiac autonomic reflex tests or severe abnormalities in orthostatic blood pressure (T2D N+ group)
6. Signed the informed consent.
7. Not defined by the exclusion criteria.

Exclusion Criteria:

1. Severe decreased liver function (Alanin amino-transaminase (ALAT) >250 U/l, Gamma-Glutamyltransferase (GGT) >150 U/l).
2. Moderate to severe kidney dysfunction, estimated Glomerular Filtration Rate (eGFR) <15 mmol/L/1,73m2.
3. Pregnancy or breast feeding.
4. Active malignancy or terminal ill.
5. Previous chemotherapy or immunomodulating treatment
6. Known severe vitamin deficiency
7. Current or previous alcohol- or drug abuse.
8. Not being able to understand Danish written and/or verbally.
9. Terms according to investigators judgement that makes subjects unsuitable to participate including lack of ability to understand and comply with instructions and/or reduced physical ability, limiting the ability to participate in the examinations.
10. Participating in other clinical studies utilizing experimental treatment or medication.
11. Subjects with pathologic fractures (defined as fractures due to local tumors, tumor-like lesions, or focal demineralization as visualized on radiographs).
12. Primary hyperparathyroidism, Paget's disease and other metabolic bone diseases, uncontrolled thyrotoxicosis, celiac disease not controlled by diet, known hypogonadism, severe COPD, hypopituitarism, Cushing's disease.
13. Fracture < 6 month ago
14. Initiation of antiresorptive or bone anabolic drugs <12 months ago to ensure stable bone turnover markers.
15. History of fractures following the diagnosis of diabetes (T2D F-/N- and T2D N+ groups).
16. History of peripheral or autonomic neuropathy defined by cardiac autonomic reflex tests or severe abnormalities in orthostatic blood pressure (T2D F-/N- group).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: T2D with and without fractures and neuropathy.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-02-24 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Evaluation of differences in bone microarchitecture between T2D patients with and without previous fractures assessed by HRpQCT. | Through study completion, estimated 3.5 years
  Bone microarchitecture is a composite outcome assessed by HRpQCT at radius and tibia: Total volumetric mineral density, Trabecular volumetric mineral density, Cortical volumetric mineral density, Trabecular number, Trabecular thickness, Cortical thickness, Trabecular separation, Cortical porosity, bone stiffness and failure load.
Differences in Bone material strength index (BMSi) between T2D patients with and without previous fractures measured by microindentation. | Through study completion, estimated 3.5 years
Evaluation of differences in bone turnover markers between T2D patients with and without previous fractures by biochemical analysis of different bone markers (CTX, P1NP, osteocalcin (OC), ucOC, sclerostin, osteoglycin and osteopontin). | Through study completion, estimated 3.5 years

SECONDARY OUTCOMES:
The impact of autonomic neuropathy on bone microarchitecture in T2D assessed by HR-pQCT. | Through study completion, estimated 3.5 years
  Compare bone microarchitectural parameters (assessed by HR-pQCT) in T2D patients with and without autonomic neuropathy (assessed by CAN-score from Vagus™ device, COMPASS31-score, intraepidermal nerve fiber density, orthostatic BP and ECG).
The impact of autonomic neuropathy on bone material strength in T2D assessed by microindentation. | Through study completion, estimated 3.5 years
  Compare bone material strength (assessed by microindentation) in T2D patients with and without autonomic neuropathy (assessed by CAN-score from Vagus™ device, COMPASS31-score, intraepidermal nerve fiber density, orthostatic BP and ECG).
The impact of autonomic neuropathy on bone turnover markers in T2D. | Through study completion, estimated 3.5 years
  Compare bone turnover markers in T2D patients with and without autonomic neuropathy (assessed by CAN-score from Vagus™ device, COMPASS31-score, intraepidermal nerve fiber density, orthostatic BP and ECG)
The impact of peripheral neuropathy on bone microarchitecture in T2D assessed by HR-pQCT. | Through study completion, estimated 3.5 years
  Compare bone microarchitectural parameters (assessed by HR-pQCT) in T2D patients with and without peripheral neuropathy (assessed by MNSI, PTT, QST, sural nerve conduction study and intraepidermal nerve fiber density)
The impact of peripheral neuropathy on bone material strength in T2D assessed by microindentation. | Through study completion, estimated 3.5 years
  Compare bone material strength (assessed by microindentation) in T2D patients with and without peripheral neuropathy (assessed by MNSI, PTT, QST, sural nerve conduction study and intraepidermal nerve fiber density)
The impact of peripheral neuropathy on bone turnover markers in T2D. | Through study completion, estimated 3.5 years
  Compare bone turnover markers in T2D patients with and without peripheral neuropathy (assessed by MNSI, PTT, QST, sural nerve conduction study and intraepidermal nerve fiber density).
Compare postural control between T2D patients with and without fractures assessed by force platform. | Through study completion, estimated 3.5 years
Compare postural control between T2D patients with and without peripheral/autonomic neuropathy. | Through study completion, estimated 3.5 years
  Neuropathy assessed by PTT, QST, sural nerve conduction study, skin biopsies, COMPASS-31, MNSI and Vagus device. Postural control assessed by force platform.
Compare muscle mass and strength in T2D patients with and without fractures | Through study completion, estimated 3.5 years
  Compare muscle mass (assessed by DXA scan) and muscle strength (assessed by hand grip, leg extension strength and functional tests) in T2D patients with and without fractures.
Compare muscle mass and strength in T2D patients with and without neuropathy | Through study completion, estimated 3.5 years
  Compare muscle mass (assessed by DXA scan) and muscle strength (assessed by hand grip, leg extension strength and functional tests) in T2D patients with and without neuropathy (assessed by PTT, QST, sural nerve conduction study, skin biopsies, COMPASS-31, MNSI and Vagus device).

OTHER OUTCOMES:
Co-existence of peripheral and autonomic neuropathy | Through study completion, estimated 3.5 years
  Presence of autonomic neuropathy (assessed by CAN-score from Vagus™ device, COMPASS31-score, intraepidermal nerve fiber density, orthostatic BP and ECG) will be compared with presence of peripheral neuropathy (assessed by PTT, QST, sural nerve conduction test and intraepidermal nerve fiber density) in T2D.
The impact of insulin resistance (assessed by HOMA-IR and -%B) on bone microarchitecture (assessed by HR-pQCT) in T2D. | Through study completion, estimated 3.5 years
The impact of insulin resistance (assessed by HOMA-IR and -%B) on bone material strength (assessed by microindentation) in T2D. | Through study completion, estimated 3.5 years
The impact of insulin resistance (assessed by HOMA-IR and -%B) on bone turnover markers in T2D. | Through study completion, estimated 3.5 years
The correlation between levels of Advanced Glycation End Products (AGEs) (assessed by skin autofluorescence) and bone material strength (assessed by microindentation). | Through study completion, estimated 3.5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Steno Diabetes Center Nordjylland, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Potential analysis of skin biopsies in external lab

DOCUMENTS (1):
  • Study Protocol (2023-06-27): https://cdn.clinicaltrials.gov/large-docs/43/NCT05642143/Prot_002.pdf